CLINICAL TRIAL: NCT04083898
Title: A Phase I/II Trial of Isatuximab, Bendamustine, and Prednisone in Refractory Multiple Myeloma
Brief Title: Isatuximab, Bendamustine, and Prednisone in Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision made to not move forward with Phase II portion of trial
Sponsor: Washington University School of Medicine (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201910194
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Bendamustine Hydrochloride; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Phase I Dose Level 1: Isatuximab + Bendamustine + Prednisone (Experimental): -Isatuximab (10 mg/kg) on Days 1, 8, 15, and 22 during Cycle 1 and on Days 1 and 15 of subsequent cycles. Bendamustine (50 mg/m^2) will be administered on Days 1 and 2 and prednisone (60 mg) will be administered on Days 1 through 4 of each cycle.
  Interventions: Biological: Isatuximab; Drug: Bendamustine; Drug: Prednisone
- Phase I Dose Level 2: Isatuximab + Bendamustine + Prednisone (Experimental): -Isatuximab (10 mg/kg) on Days 1, 8, 15, and 22 during Cycle 1 and on Days 1 and 15 of subsequent cycles. Bendamustine (75 mg/m^2) will be administered on Days 1 and 2 and prednisone (60 mg) will be administered on Days 1 through 4 of each cycle.
  Interventions: Biological: Isatuximab; Drug: Bendamustine; Drug: Prednisone
- Phase I Dose Level 3: Isatuximab + Bendamustine + Prednisone (Experimental): -Isatuximab (10 mg/kg) on Days 1, 8, 15, and 22 during Cycle 1 and on Days 1 and 15 of subsequent cycles. Bendamustine (100 mg/m^2) will be administered on Days 1 and 2 and prednisone (60 mg) will be administered on Days 1 through 4 of each cycle.
  Interventions: Biological: Isatuximab; Drug: Bendamustine; Drug: Prednisone
- Phase II: Isatuximab + Bendamustine + Prednisone (Experimental): -Isatuximab (10 mg/kg) on Days 1, 8, 15, and 22 during Cycle 1 and on Days 1 and 15 of subsequent cycles. Bendamustine (dose determined in Phase I portion of study) will be administered on Days 1 and 2 and prednisone (60 mg) will be administered on Days 1 through 4 of each cycle.
  Interventions: Biological: Isatuximab; Drug: Bendamustine; Drug: Prednisone

INTERVENTIONS:
Biological: Isatuximab — Isatuximab will be administered on a 28-day cycle
Drug: Bendamustine — Bendamustine will be administered on a 28-day cycle as follows
  Other Names: Bendeka; Treanda
Drug: Prednisone — Prednisone will be administered on a 28-day cycle as follows
  Other Names: Deltasone; Rayos; Prednisone Intensol

SUMMARY:
Isatuximab targets and kills CD38-positive myeloma cells in manner similar to rituximab's mechanism of action on CD20-positive lymphoma cells. Based on the synergy between rituximab and bendamustine, as well as the established clinical efficacy of bendamustine and isatuximab as single agents for multiple myeloma, the logical next step is to combine isatuximab with bendamustine and prednisone. Due to lack of effective therapies in refractory multiple myeloma, herein the investigators propose studying this novel combination in this population, in order to address a significant unmet need. The aim of the investigators is to first determine the maximal tolerated dose of the combination in participants with relapsed/refractory myeloma and then to establish the efficacy of this novel combination.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma with a measurable disease parameter at time of screening. A measurable disease parameter is defined as one or more of the following:

  * Serum monoclonal protein ≥ 0.5 g/dL
  * 24 hour urine monoclonal protein ≥ 200 mg/24 hour
  * Serum free light chain ratio > 5x normal ratio with an absolute difference of 10mg/dL between the involved and uninvolved free light chain
  * Soft tissue plasmacytoma ≥ 2 cm measurable by either physical examination and/or applicable radiographs (e.g. MRI, CT, etc.)
  * Bone marrow plasma cells ≥ 30%
* Triple-class-refractory disease defined as both of the following:

  * Previously received treatment with a proteasome inhibitor, an immunomodulatory drug, and daratumumab, in combination or as single-agents.
  * Refractory (defined per IMWG Consensus Criteria as disease that is nonresponsive while on therapy, or progresses within 60 days of last dose) to most recent therapy.
* At least 6 weeks from the last treatment with daratumumab to the first study treatment
* At least 18 years of age.
* Performance status of ECOG ≤ 2 Note: Participants with lower performance status based solely on bone pain secondary to multiple myeloma will be eligible.
* Normal bone marrow and organ function as defined as ALL of the following:

  * Absolute neutrophil count ≥ 1500/mm3
  * Platelets ≥ 75,000/mm^3 (transfusions not permitted within 7 days of screening)
  * ALT (SGPT) and AST (SGOT) < 3.5 x the upper limit of the institutional normal value (ULN).
  * Total bilirubin ≤ 2.0 x mg/dL.
  * Creatinine clearance > 30 ml/min using Cockcroft-Gault formula
* Females of childbearing potential (FCBP) must agree to refrain from becoming pregnant while on study drug and for 3 months after discontinuation from study drug, and must agree to use adequate contraception including hormonal contraception, (e.g. birth control pills, etc.), barrier method contraception (e.g. condoms), or abstinence during that time frame. Men engaging in sexual intercourse with a FCBP must agree to use adequate contraception including hormonal contraception, (e.g. birth control pills, etc), barrier method contraception (e.g. condoms), or abstinence while on study drug and for 3 months after discontinuation from study drug
* Ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Prior exposure to isatuximab or bendamustine
* History of plasma cell leukemia or MM CNS involvement.
* Receiving renal replacement therapy, hemodialysis, or peritoneal dialysis.
* Diagnosed with another concurrent malignancy requiring treatment.
* Active hepatitis A, B, or C.
* Known intolerance to infused protein products, sucrose, histidine, polysorbate 80 or known hypersensitivity to any of the components of study therapy.
* Receiving any other investigational agents within 14 days prior to enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of regimen (Phase I only) | Completion of first cycle of treatment for all participants enrolled in Phase I portion (estimated to be 9 months)
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 participants of a cohort (of 2 to 6 participants) experience dose limiting toxicity (DLT) during the first cycle of treatment. Dose escalation will proceed until the MTD has been reached or until the maximum dose of each drug is tested (Dose Level 3). If no more than 1 DLT is observed at dose levels 1, 2 and 3, level 3 will be declared the recommended phase II dose (RP2D) and the MTD will remain undefined.
Overall response rate (ORR) (Phase II only) | 6 months
  -ORR defined as the proportion of patients meeting the criteria for partial response, very good partial response, complete response, or stringent complete response per IMWG 2016 response criteria.

SECONDARY OUTCOMES:
Number of adverse events experienced by participants (Phase I and Phase II) | From start of treatment through 30 days after completion of treatment or initiation of new anti-myeloma therapy, whichever occurs first (estimated to be 7 months)
  Participants will be evaluated for toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute (NCI) version 5.0.
Progression-free survival (PFS) (Phase II only) | Up to 5 years after removal from study (estimated to be 5 years and 6 months)
  Progression-free survival (PFS) will be defined as time from Cycle 1 Day 1 to disease progression or relapse. Any patient who expires, withdraws, or is lost to follow-up prior to disease progression or relapse will be censored at last follow-up. Patients who are removed from study therapy prior to progression or relapse will be censored at the time of initiation of subsequent anti-myeloma treatment.
Overall survival (OS) (Phase II only) | Up to 5 years after removal from study (estimated to be 5 years and 6 months)
  Overall survival (OS) will be defined as time from Cycle 1 Day 1 to death due to any causes. Patients who are alive at the time of data analyses will be censored on the last known alive date. Patients who are removed from study therapy prior death will be censored at the time of initiation of subsequent anti-myeloma treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldsmith SR, Slade MJ, Fiala M, Harding M, Crees ZD, Schroeder MA, Stockerl-Goldstein K, Vij R. A phase Ib trial of isatuximab, bendamustine, and prednisone in relapsed/refractory multiple myeloma. Ann Hematol. 2024 Nov;103(11):4557-4565. doi: 10.1007/s00277-024-05975-7. Epub 2024 Sep 4. PMID 39227452
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu